CLINICAL TRIAL: NCT02631460
Title: A Randomized Phase II Study of S1 Plus Carboplatin Followed by Maintenance S1versus Pemetrexed Plus Carboplatin Followed by Maintenance Pemetrexed in Patients With EGFR Wild Type Stage IIIB or IV Nonsquamous Non-Small-Cell Lung Cancer
Brief Title: S1 vs.Pemetrexed Plus Carboplatin in Patients With EGFR Wild Type Stage IIIB or IV Nonsquamous NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5010-2015023
Record Dates: First submitted 2015-12-12; First posted 2015-12-16 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: NSCLC
MeSH Terms: interventions — S 1 (combination); Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- S1 and Carboplatin (Experimental): S1 80-120 mg/d+Carboplatin AUC=5 Patients without progression received maintenance until disease progression with S1
  Interventions: Drug: S1 80-120 mg/d; Drug: carboplatin AUC=5
- pemetrexed and Carboplatin (Active Comparator): pemetrexed 500 mg/m2+ Carboplatin AUC=5 Patients without progression received maintenance until disease progression with pemetrexed
  Interventions: Drug: pemetrexed 500 mg/m2; Drug: carboplatin AUC=5

INTERVENTIONS:
Drug: S1 80-120 mg/d — d1, every 3 weeks
  Arms: S1 and Carboplatin
Drug: pemetrexed 500 mg/m2 — d1, every 3 weeks
  Arms: pemetrexed and Carboplatin
Drug: carboplatin AUC=5 — d1, every 3 weeks

SUMMARY:
This study compared the efficacy and safety of S1 plus carboplatin (C) followed by S1 with pemetrexed plus carboplatin (C) followed by pemetrexed in patients with epidermal growth factor receptor (EGFR) wild type advanced nonsquamous non-small-cell lung cancer (NSCLC).Patients with previously untreated EGFR wild type stage IIIB or IV nonsquamous NSCLC and Eastern Cooperative Oncology Group performance status of 0 to 1 were randomly assigned to receive pemetrexed 500 mg/m2 or S1（80-120 mg/d）combined with carboplatin area under the curve (AUC) 5 every 3 weeks for up to four cycles. Eligible patients received maintenance until disease progression: pemetrexed or S1. The primary end point of this non-inferiority study was progression free survival（PFS）

ELIGIBILITY:
Inclusion Criteria:

1. Chemotherapy-naive patients with histologically or cytologically confirmed nonsquamous NSCLC, classified as stage IIIB not amenable to curative treatment or stage IV; EGFR wild type.
2. At least one unidimensionally measurable lesion according to the Response Evaluation Criteria in Solid Tumors
3. Eastern Cooperative Oncology Group performance status of 0 or 1
4. 18 <age<75 years
5. Patients had adequate bone marrow reserve and organ function.
6. Prior radiation therapy was permitted if it was completed at least 4 weeks before study treatment and patients had fully recovered from its acute effects
7. Written informed consent was obtained directly from every patient
8. Estimated life expectancy of at least 12 weeks.
9. Patient compliance and geographic proximity that allow adequate follow up.
10. Male and female patients with reproductive potential must use an approved contraceptive method, if appropriate during and for 3 months after the study. Women with childbearing potential must have a negative serum pregnancy test within 7 days prior to study enrollment.

Exclusion Criteria:

1. Brain metastasis associated with central nervous symptoms (patients were eligible if symptoms were controlled by steroids or other treatments);
2. Serious infections or other serious complications.
3. Uncontrolled third-space fluid retention before study entry. unable to interrupt aspirin and other nonsteroidal anti-inflammatory drugs or if they were unable or unwilling to take folic acid, vitamin B12, or corticosteroids
4. Have a prior malignancy other than NSCLC, carcinoma in situ of the cervix, or nonmelanoma skin cancer, unless that prior malignancy was diagnosed and definitively treated at least 5 years previously with no subsequent evidence of recurrence.
5. Pregnant or breast feeding.
6. A distinct history of drug allergies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival(PFS) | 3 years

SECONDARY OUTCOMES:
Overall survival(OS) | 4 years
Disease control rate(DCR) | 3 years
Health-related quality of life | 3 years
Number of Participants with Adverse Events | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Yan Huang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun yat-sen University Cancer Center, Guangzhou, Guangdong, China